CLINICAL TRIAL: NCT01771562
Title: Assessment of Risk Factors of Nutritional and Metabolic Disorders in Children and Adolescent Receiving or Not Antiretroviral Treatment : Growing up With HIV in Senegal
Brief Title: Nutritional and Metabolic Disorders in HIV Infected Children and Adolescent
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 12279 MAGGSEN
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: HIV-1
Keywords: HIV-1; Child; Adolescent; Growth; Lipodystrophy; ARV treatment; Senegal
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Plasma, blood cells and urine samples to be retained
Oversight: Data Monitoring Committee: No

SUMMARY:
The advent of highly active antiretroviral treatment has resulted in the survival into adolescence of an increasing proportion of infants and children with perinatal HIV infection in Senegal. However, the transformation of HIV into a chronic disease needing lifelong antiretroviral treatment (ART) raises new challenges, among others related to a disturbance of glucose metabolism, lipid abnormalities, in addition to the potential effects on children's growth and puberty. Little is known on nutritional and metabolic changes in HIV-infected children on ART in Africa, while implementation of the latest WHO recommendations should eventually lead to an increase in the number of children on ART in this region. Moreover, bio-clinical evolution of untreated children is poorly documented in the African context. It therefore urgently needed to institute a cohort study to evaluate, in the long term, the impact of HIV infection and/or ART on nutritional and metabolic disorders and to characterize the risk factors of their occurrence in children and adolescents infected as they move through adolescent into adulthood.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Age equal or above 2 years and bellow 16 years
* Follow-up in the participating site
* Informed consent signed by at least on of the parents or legal guardian who is aware of the child's HIV status

Exclusion Criteria:

* HIV-2 or HIV-1+2 infection
* children represented by a legal guardian who is not informed about the child's HIV status
* Unable to comply with study requirements or procedures according to the investigator's opinion

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: HIV-1 infected individuals age between 2 ans 16 years
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of delayed growth | Baseline
  Delayed growth is defined by height for age < -2 z-scores, wasting (%) by weight-for height < -2 z-scores and/or BMI-age < -2 z-scores
Prevalence of delayed puberty | Baseline
  Delayed puberty is assessed by age of entry into puberty and the age of transition to different Tanner staging
Prevalence of lipodystrophy | Baseline
  Lipodystrophy (lipoatrophy, lipohypertrophy, combined forms) is defined by direct observation and by joint analysis of anthropometric measures associated with fat tissue index and lean tissue index measured by electrical bio-impedancemetry
Prevalence of blood lipids ans glucose abnormalities | Baseline
  Measurement of blood glucose, total cholesterol, HDL, LDL and triglycerides
Incidence of delayed growth | Annually for 3 years from the anniversary date of the study
  Delayed growth is defined by height for age < -2 z-scores, wasting (%) by weight-for height < -2 z-scores and/or BMI-age < -2 z-scores
Incidence of delayed puberty | Annually for 3 years from the anniversary date of the study
  Assessed by age of entry into puberty and the age of transition to a different Tanner stage
Incidence of lipodystrophy | Annually for 3 years from the anniversary date of the study
  defined by direct observation and by joint analysis of anthropometric measures associated with changes in fat tissue index and lean tissue index measured by electrical bio-impedancemetry
Incidence of blood lipid and glucose abnormalities | Annually for 3 years from the anniversary date of the study
  Repeated measurement of blood glucose, total cholesterol, HDL, LDL and triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Msellati, MD, Principal Investigator — IRD : French Research Institute for Development; Haby Sy Signate, MD, Principal Investigator — Hôpital d'Enfant Albert Royer, Dakar, Senegal; Ngagne Mbaye, MD, Principal Investigator — Hôpital Roi Baudoin, Guédiawaye, Senegal
Locations (2):
- Senegal (2):
  - Hôpital d'enfant Albert Royer, Dakar
  - Hôpital Roi Baudoin, Guédiawaye

REFERENCES:
- [Derived] Cames C, Pascal L, Ba A, Mbodj H, Ouattara B, Diallo NF, Msellati P, Mbaye N, Sy Signate H, Blanche S, Diack A; MAGGSEN Cohort Study Group. Low prevalence of lipodystrophy in HIV-infected Senegalese children on long-term antiretroviral treatment: the ANRS 12279 MAGGSEN Pediatric Cohort Study. BMC Infect Dis. 2018 Aug 6;18(1):374. doi: 10.1186/s12879-018-3282-7. PMID 30081838
- [Derived] Cames C, Varloteaux M, Have NN, Diom AB, Msellati P, Mbaye N, Mbodj H, Sy Signate H, Diack A; ANRS 12279 MAGGSEN Cohort Study Group. Acceptability of Outpatient Ready-To-Use Food-Based Protocols in HIV-Infected Senegalese Children and Adolescents Within the MAGGSEN Cohort Study. Food Nutr Bull. 2017 Mar;38(1):27-36. doi: 10.1177/0379572116679053. Epub 2016 Nov 23. PMID 27881690
- See also: Sponsor website — http://www.anrs.fr